CLINICAL TRIAL: NCT03111680
Title: Healthy Families: a Cluster Randomized Study to Change Obesity in Public Housing
Brief Title: Healthy Families to Change Obesity in Public Housing Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Deborah Bowen, Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: U48DP001922 (NIH)
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Milieu Therapy

STUDY DESIGN:
Intervention Model Description: this was a cluster randomized trial, with housing developments randomized to intervention or control
Who Masked: Care Provider, Investigator
Masking Description: people collecting data were unaware of study condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): this arm received an environmental intervention to make healthy eating and activity easier for residents
  Interventions: Other: environmental intervention
- control (No Intervention): the control participants received no interventions

INTERVENTIONS:
Other: environmental intervention — a multi component environmental intervention
  Arms: intervention

SUMMARY:
This is a cluster randomized study of an environmental level intervention to improve nutrition and physical activity, among public housing residents. Followup was one year post baseline

DETAILED DESCRIPTION:
Purpose and design The purpose of this study was to test the effects of a environmental-level package of interventions on public housing residents' obesity and obesity-related behaviors. The design of the study and its intervention have been previously published . Simply, this was a cluster randomized trial, with public housing developments (PHDs) serving as the unit of randomization and analysis. This document describes the patterns of change in the main behavioral and weight outcomes for adult women before and after the intervention.

Participants Public housing in Boston is administered by the Boston Housing Authority (BHA), a public agency that provides subsidized housing to low- and moderate-income individuals and families, disabled individuals, and elderly individuals. There are 64 public housing developments, 37 are designated as elderly/disabled developments and 27 are designated as family developments. Approximately 27,000 people are housed under the public housing program.

Family (vs. elderly) designated PHDs with more than 200 residents which were not undergoing renovations requiring residents to move out of the development for a period of time in the City of Boston were eligible to participate in this study (n=24). The investigators recruited 10 developments to participate in the Healthy Families study; 5 serving as intervention PHDs and 5 serving as control PHDs. PHDs were randomly assigned to either condition, in matched pairs for size of development and existence of health activities in the development. PHDs randomized to the intervention group received all intervention components (see Intervention section below) and developments randomized to the control group did not receive any intervention components.

Data collection In both intervention and control group PHDs, a randomly sampled group of female residents and their daughters ages 8-16 were recruited into an evaluation cohort to examine study outcomes. The investigators selected mothers because in the family developments over 80% of heads of household (per aggregate data compiled from tenant agreements) were women. The investigators selected daughters aged 8-15 as development of obesity often occurs during this time period for females. To be eligible for this study, participants were required to be female, age 18-72, live in one of the recruited PHD, and planning to remain so for two years, had responsibility for a girl age 8-15 (also living in the public housing residence), were English or Spanish speaking, and were able to make changes to their diet and physical activity habits if desired. Exclusion criteria included: the adult was not able to complete the survey tools or was not interested in participating. All study materials were available and used in both English and Spanish.

Survey assistants approached randomly selected apartment units within each of the 10 housing developments. Using a standardized protocol, survey assistants assessed individual's interest in participating and eligibility. If interested and eligible, the participant provided their written informed consent to participate, girls aged 12-15 provided written assent, and girls aged 8-11 gave verbal assent. The survey assistant then administered the baseline survey and recorded the (adult) participant's responses. After completing the survey, the women and girl's height and weight were measured and recorded. Project staff returned to re-assess the original evaluation cohort at one- year follow-up.

Measures Baseline survey. Dietary intake is difficult and time consuming to measure, and so in the interest of minimizing participant burden we decided to measure key single behaviors related to obesity for which there were existing measures. Following evidenced-based guidelines for health promotion and weight management, we assessed three nutrition behaviors: fruits and vegetables ("How many servings of fruits and vegetables do you eat each day?" with 12 responses ranging from 0 to 11 or more, which was prefaced with pictures representing portion sizes); soda ("How often do you drink soft drinks or soda pop (regular or diet)?" with 6 responses ranging from never to 2 or more times per day); mindless eating ("How often do you eat food (meals or snacks) while doing another activity, for example, watching TV, working at a computer, reading, driving, playing video games?" with 5 responses ranging from never to always). The same measurement difficulties exist for physical activity, and so investigators used the same strategy to select key single items that have been used before in research studies and compared well with longer measures. We assessed physical activity in the form of walking for leisure, transport, or exercise during the past week with the following question: "During the last 7 days, on how many days did you walk for at least 10 minutes at a time in your neighborhood?" with responses ranging from no walking for more than 10 minutes at a time or the option to fill in number of days per week and number of minutes per day. Number of days/week was multiplied by minutes/day to calculate minutes of walking per week. To assess walking on a typical day, we then asked: "On a typical day how many minutes do you walk in your neighborhood?" with the option to fill in minutes per day. Finally, the survey assistant measured the height and weight of both the mother and daughter using a scale. This was used to calculate body mass index (BMI, kg/m2). Both body weight and survey variables were planned to occur annually for the duration of the study.

Participants completed standard questions about socio-demographics (e.g., age, race/ethnicity, highest level of education completed, self-rated health), psychosocial, and behavioral variables. To assess self-efficacy to eat more healthfully, surveys asked "On a scale of 0 to 10, how sure are you that you will eat less sugar and fat during the next year?" with 11 responses ranging from 0 (not sure) to 10 (very sure).

Intervention The Healthy Families intervention was developed using the conceptual model depicting the mother-daughter pairs who are at the center of our intervention surrounded by three main environmental-level categories of influence: community, organizational, and consumer nutrition and physical activity environments. The main emphasis of the model is on various environmental influences, with individual-level factors, socio-demographics and psychosocial factors, influencing eating and physical activity patterns. Healthy Families contained multiple intervention components: lay health advisors, health screenings, walking groups, nutrition and cooking demonstrations, healthy purchasing options, and neighborhood resource maps. Investigators chose these components to comprise our intervention since they could be implemented within a short period of time, could be sustained by the developments at the conclusion of our project, and were built on research already conducted by the Partners in Health and Housing=Prevention Research Center.

Lay Health Advisors. The intervention components were coordinated by residents of public housing who had completed a 14-week training in community health outreach, a long-standing program (12+ years) provided by the PHH-PRC. Upon completion, these lay health advisors complete a six month paid internship in their public housing development, distributing health information on a variety of topics of concern to residents and helping to link residents to neighborhood health- and clinical-related resources. From the pool of approximately 100 lay health advisors, a subset was selected to be trained in obesity-specific knowledge and procedures to serve in the Healthy Families intervention. They completed an additional 3-day training covering research processes (e.g., protecting participant privacy), study-specific protocols, and obesity management (e.g., health implications of obesity, effective approaches to supporting weight loss) and passed a post-training assessment to demonstrate their knowledge. Upon completion, these trained residents, called Healthy Living Advocates (HLAs) (n=5), served to coordinate the Healthy Family activities, described below, in the 5 intervention developments.

Health screenings. Screening for risk factors for chronic disease is one of the most widely used strategies to prevent mortality and morbidity for chronic disease in modern industrialized countries. Identification of risk factors, measured in blood or other body fluids, or by body function, like blood pressure, offers information about a person's overall risk for development of chronic diseases, like cardiovascular disease and diabetes. Among public housing residents, we found in previous work that both rates of participation in screenings and the rates of positive screens for chronic disease was high among residents when the screenings were held inside the housing developments. Therefore, the study offered monthly screenings for blood pressure, smoking, and diabetes risk for individuals to learn about their chronic disease risk and be referred to a program within the Healthy Families intervention, to their own provider, or given information about how to obtain a provider if they did not have one. Due to expanded public insurance options, 94-97% of non-elderly adults in Massachusetts had health insurance at the time of this project, removing this classic barrier to care. The screenings were 3-4 hours in duration, held in a shared space in the development, were advertised for 2 weeks prior, and were administered by research study staff. HLAs attended all screenings to assist with linking residents to the primary care system as needed.

Access to healthy food. Increasing access to healthy foods is a key component of improving the food environment, yet, adding supermarkets or changing the existing store resources (e.g., adding refrigerated units to accommodate fruits and vegetables) can takes years to perform and are often expensive. Additional options, such as farmer's markets and urban gardening, can be limited by their seasonal nature and may have differential patterns of use in different areas of the U.S. To provide immediate, affordable, and easy access to healthy choices, we selected providing access in the form of a van (Fresh Truck) that sold fruits and vegetables to residents of public housing. The van visited each intervention housing development weekly. HLAs at each development promoted the van's offerings and were present while the Fresh Truck was parked on-site.

Walking groups. Research suggests that the built environment is a powerful influence on behaviors. Significant environmental barriers to walking, particularly among multi-cultural low-income women, have been well-documented and include lack of sense of safety and lack of places to exercise. Pilot work indicates that walking groups are well-accepted by public housing residents, with about 20% of residents participating across 4 housing complexes, reporting self-reported increases in days of walking and social cohesion. Walking groups were held weekly, with HLAs serving as walk group leaders and promoting the groups in the developments via flyers and word of mouth.

Cooking demonstration. Numerous successful multi-component interventions with the aim of reducing overweight and obesity have used cooking demonstrations as part of their programming. These cooking demonstrations offered residents the opportunity to obtain nutrition education as well as to shape social norms around healthful food practices among friends/family/neighbors. A common theme of our cooking demonstrations was tailoring recipes to fit the targeted cultural context. Prior to the Healthy Families project, nearly all residents and management at targeted developments reported a desire to bring cooking classes to their neighborhoods as they were thought of as family-friendly activities and positive social functions in which neighbors could get together and work towards a common goal. The cooking demonstrations were held four times per development, led by a Registered Dietitian, and promoted beforehand by the HLAs using flyers and word of mouth, as well as via social media. The dietitian compiled a number of culturally diverse recipes which included foods that were available for purchase from the Fresh Food Truck and were SNAP eligible and WIC approved. At each demonstration, the dietitian prepared two recipes and provided nutrition education on a number of topics such as whole grains and sodium reduction.

Resource maps. Maps listing local health related resources (such as local gyms, walking parks, and healthy buying and eating establishments) were made available to development leaders and to all interested participants at health screenings, food van session, walking groups, and cooking demonstrations.

ELIGIBILITY:
Inclusion Criteria:

* residing in public housing able to read spanish or english mother of a child aged 6-17

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 211 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
healthy eating | in the last three months
  fruit and vegetable servings per day
healthy physical activity | in the last three months
  time spent doing moderate physcial activity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quintiliani LM, DeBiasse MA, Branco JM, Bhosrekar SG, Rorie JA, Bowen DJ. Enhancing physical and social environments to reduce obesity among public housing residents: rationale, trial design, and baseline data for the Healthy Families study. Contemp Clin Trials. 2014 Nov;39(2):201-10. doi: 10.1016/j.cct.2014.08.005. Epub 2014 Aug 17. PMID 25139728